CLINICAL TRIAL: NCT03468023
Title: Short vs Long Arm Cast for Distal Radius Fractures: the Verona Trial. Randomized Clinical Trial to Assess the Efficacy of Short Arm Cast Versus Long Arm Cast in Conservative Management of Distal Radius Fractures
Brief Title: Short vs Long Arm Cast for Distal Radius Fractures: the Verona Trial
Acronym: SLA-Ver
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Tommaso Maluta, Principal Investigator, Azienda Ospedaliera Universitaria Integrata Verona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1165CESC; 1166CESC (Registry Identifier: Comitato Etico per la sperimentazione clinica delle province di Verona e Rovigo)
Record Dates: First submitted 2018-03-11; First posted 2018-03-16 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Radius Fracture Distal
Keywords: Cast treatment; above-elbow cast; below-elbow cast; long arm cast; short arm cast
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Intervention Model Description: Non-inferiority trial aimed at comparing the non inferiority of a short arm cast (below elbow cast) as opposed to a long arm cast (below elbow cast) in terms of fracture reduction maintenance ratio.
  The sample size was selected as the highest required to test all non-inferiority thresholds and considering a drop-out percentage of 15%. Continuous values of all radiological parameters were used in order to keep results objective and reproducible.
  At the end of recruitment observed drop-out percentage was 26%.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short arm cast (Experimental): Patient treated with below-elbow cast
  Interventions: Procedure: Short arm cast
- Long arm cast (Active Comparator): Patients treated with above-elbow cast
  Interventions: Procedure: Long arm cast

INTERVENTIONS:
Procedure: Short arm cast — Application of a below-elbow cast
  Other Names: below-elbow cast; antebrachio-metacarpal cast
  Arms: Short arm cast
Procedure: Long arm cast — Application of an above-elbow cast
  Other Names: above-elbow cast; brachio-metacarpal cast
  Arms: Long arm cast

SUMMARY:
This study prospectively compares the performance of an above-elbow cast (long arm cast) and a below-elbow cast (short arm cast) to maintain reduction in conservatively managed distal radius fractures.

DETAILED DESCRIPTION:
The choice of cast length in conservative management of distal radius fractures still represents a much debated controversy. Classic teaching was to immobilize the elbow to reduce risk of secondary displacement; however, short arm casts are felt to be equally effective with less complications and higher patient comfort. There is currently no conclusive evidence for or against immobilization of the elbow in patients treated with cast immobilization.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of distal radius fracture
* Indication to conservative treatment
* Need for manipulation to reduce fracture

Exclusion Criteria:

* Open fractures
* Existence of any skin lesion or wound that would impair cast treatment
* Neurovascular deficits
* Bilateral fractures
* Association with any other fracture of the homolateral arm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2020-03-28 (Actual)

PRIMARY OUTCOMES:
Secondary displacement ratio | 35 days
  Percentage of fractures that displace during treatment as subjectively assessed on radiographs by investigators.
Variation of radial length | 35 days
  Difference between radial length values as objectively measured on postreduction radiographs and endtreatment radiographs.
Variation of radial inclination | 35 days
  Difference between radial inclination values as objectively measured on postreduction radiographs and endtreatment radiographs.
Variation of volar tilt | 35 days
  Difference between volar tilt vaues as objectively measured on postreduction radiographs and endtreatment radiographs.

SECONDARY OUTCOMES:
Post-treatment elbow range of motion (ROM) | 35 days
  Degrees of extension, flexion, pronation and supination of the elbow measured at the end of the treatment.
DASH score | 35 days
  Disability of Arm, Shoulder and Hand score measured at the end of the treatment relating to patient's comfort during treatment.
SF-12 | 35 days
  Short Form 12 health questionnaire administered at the end of the treatment relating to patient's quality of life during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Tommaso Maluta, MD, Study Director — Azienda Ospedaliera Universitaria Integrata Verona; Giovanni Dib, MD, Principal Investigator — Azienda Ospedaliera Universitaria Integrata Verona; Matteo Cengarle, MD, Principal Investigator — Azienda Ospedaliera Universitaria Integrata Verona; Alice Bernasconi, DR, Principal Investigator — Azienda Ospedaliera Universitaria Integrata Verona; Franco Lavini, MD, Principal Investigator — Azienda Ospedaliera Universitaria Integrata Verona; Andrea Scalvi, MD, Study Chair — Azienda Ospedaliera Universitaria Integrata Verona; Bruno Magnan, MD, Study Chair — Azienda Ospedaliera Universitaria Integrata Verona
Locations (1):
- Ospedale Civile Maggiore Borgo Trento, Verona, Italy

REFERENCES:
- [Derived] Dib G, Maluta T, Cengarle M, Bernasconi A, Marconato G, Corain M, Magnan B. Short arm cast is as effective as long arm cast in maintaining distal radius fracture reduction: Results of the SLA-VER noninferiority trial. World J Orthop. 2022 Sep 18;13(9):802-811. doi: 10.5312/wjo.v13.i9.802. eCollection 2022 Sep 18. PMID 36189333